CLINICAL TRIAL: NCT05120726
Title: A Novel Therapeutic Treatment of Pyoderma Gangrenosum
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was closed prior to completion because of difficulties in recruiting eligible participants. Despite outreach efforts, enrollment remained insufficient to meet anticipated study endpoints.
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Alison A. Smith, Assistant Clinical Professor of Surgery, Louisiana State University Health Sciences Center in New Orleans
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB: #1579
Record Dates: First submitted 2021-09-11; First posted 2021-11-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-05

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum; EpiFix; dehydrated human amnion/chorion membrane
MeSH Terms: conditions — Pyoderma Gangrenosum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Patient's pyoderma gangrenosum wounds are treated surgically with EpiFix (dehydrated human amnion/chorion membrane). In another surgery about one week later, we will be covering the treated wounds with split-thickness skin grafts. During each surgery, we will be collecting wound samples for genetic analysis. Routine post-surgery clinic visits will be used to monitor wound healing over a 6-month period.
  Interventions: Biological: Dehydrated human amnion/chorion membrane

INTERVENTIONS:
Biological: Dehydrated human amnion/chorion membrane — Dehydrated human amnion/chorion membrane (dHACM) has been commercially available for nearly 15 years. dHACM has been shown to elute growth factors including platelet-derived growth factors, fibroblast growth factors (PDGF), fibroblast growth factors (FGF), transforming growth factor beta 1 (TGF-β1), epidermal growth factor (EGF), vascular endothelial growth factor (VEGF), and placental growth factor (PlGF). Additionally, dHACM exerts immunomodulatory effects by releasing anti-inflammatory interleukins and factors which help regulate the matrix metalloproteinase (MMP) activity. Furthermore, dHACM has also been shown to stimulate mesenchymal stem cell migration and recruitment. dHACM is routinely utilized in the management of chronic wounds including diabetic ulcer and venous ulcers.
  Other Names: EpiFix; dHACM

SUMMARY:
Pyoderma gangrenosum is a chronic debilitating ulcerative neutrophilic condition usually affecting the skin. The pathogenesis of pyoderma gangrenosum is poorly understood. Pyoderma gangrenosum has been estimated to have an incidence rate of 3-10 per million populations per year. Mortality estimates range up to 30%. The non-healing wounds present a significant social and economic burden on affected patients. We hypothesize that EpiFix (dehydrated human amnion/chorion membrane) will be beneficial in treating patients with pyoderma gangrenosum.

Potentially eligible patients will be pre-screened in clinic. The pre-screening process will include a medical history, including review of co-morbid medical problems and home medications, and a physical exam of the wounds.

The first stage of the study will involve a surgery in which the pyoderma gangrenosum wounds are going to be treated with the EpiFix. About a week later, the patient will then undergo another surgery where skin grafts will be placed on the wounds that were treated in the first surgery. In each surgery, samples of the wound will be taken, and genetic information from these samples will be studied to identify the genes that are active before and after treating the wound with EpiFix.

Routine post-surgery clinic visits will then be used to monitor the healing of the wounds and make sure that no extra medical treatment is needed. Study staff will evaluate wounds twice a week for the first two weeks, then once a week until 6 weeks. Following this, you will then be followed every 4 weeks up to 22 weeks. These visits to the clinic will include taking wound measurements, taking digital photos, asking about level of pain and evaluating development of infection. Patient consent will be obtained to take any photos.

DETAILED DESCRIPTION:
In part because of its efficacy, the number of clinical indications for dehydrated human amnion/chorion membrane (dHACM) has expanded, and a number of case reports now suggest pyoderma gangrenosum can be successfully treated with dHACM. However, the mechanisms underlying dHACM's beneficial effects is entirely unstudied. The overall goal of the proposed study is to characterize the transcriptome of a pyoderma gangrenosum wound before and after successful treatment with dHACM. We will identify certain genes or genetic pathways that are specifically targeted by treatment of a wound with dehydrated human amnion/chorion membrane (EpiFix). With this data, we hope to better understand the method by which EpiFix can specifically heal a wound. Ultimately, all this data will be used to identify specific findings that aid in the diagnosis and treatment of pyoderma gangrenosum. A previous IRB-approved study by Dr. Frank Lau at LSU and colleagues (unpublished data) investigated the use of EpiFix to treat wounds in 3 patients with pyoderma gangrenosum with success and minimal complications.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with pyoderma gangrenosum
* patients over 18 years of age

Exclusion Criteria:

* members of vulnerable populations (pregnant women and prisoners)
* patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Gene Measurements | Wound specimen are collected during each surgical intervention (over ~2 weeks)
  Identifying genes or genetic pathways that are specifically targeted by treatment of a wound with dehydrated human amnion/chorion membrane (dHACM)
Wound Size | ~6 months (post-op weeks 1, 2, 3, 4, 5, 6, 10, 14, 18, 22; +/- 2 weeks each time in case conflicts arise)
  Size of the pyoderma wound (mm)

SECONDARY OUTCOMES:
Infection | ~6 months (post-op weeks 1, 2, 3, 4, 5, 6, 10, 14, 18, 22; +/- 2 weeks each time in case conflicts arise)
  Yes/No
Pain Level | ~6 months (post-op weeks 1, 2, 3, 4, 5, 6, 10, 14, 18, 22; +/- 2 weeks each time in case conflicts arise)
  Scale (0-10) (0 = no pain, 10 = worst pain ever experienced)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Smith, MD, PhD, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (3):
- United States (3):
  - LSU Healthcare Network Clinic, Metairie, Louisiana
  - University Medical Center, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maverakis E, Marzano AV, Le ST, Callen JP, Bruggen MC, Guenova E, Dissemond J, Shinkai K, Langan SM. Pyoderma gangrenosum. Nat Rev Dis Primers. 2020 Oct 8;6(1):81. doi: 10.1038/s41572-020-0213-x. PMID 33033263
- [Background] Koob TJ, Rennert R, Zabek N, Massee M, Lim JJ, Temenoff JS, Li WW, Gurtner G. Biological properties of dehydrated human amnion/chorion composite graft: implications for chronic wound healing. Int Wound J. 2013 Oct;10(5):493-500. doi: 10.1111/iwj.12140. Epub 2013 Aug 1. PMID 23902526
- See also: EpiFix Information — http://www.mimedx.com/products/epifix/

DOCUMENTS (1):
  • Informed Consent Form (2021-03-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT05120726/ICF_000.pdf